CLINICAL TRIAL: NCT04750759
Title: A Randomized, Single Blind, Placebo-controlled, Multiple Dose, Parallel-arm Study to Investigate the Safety and Preliminary Efficacy of the Combination of Niclosamide and Camostat to Treat COVID-19 ("NICCAM")
Brief Title: Safety and Preliminary Efficacy of the Combination of Niclosamide and Camostat
Acronym: NICCAM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sub-therapeutic plasma levels of active substance
Sponsor: Charité Research Organisation GmbH (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201741
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Niclosamide; camostat

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Niclosamide + Camostat (Active Comparator): Patients will receive the combination of niclosamide chewing tablets (2000 mg, once daily) and camostat tablets (600 mg, 4-times daily) over a period of 7 days.
  Interventions: Drug: Niclosamide + Camostat
- Placebo (Placebo Comparator): Patients will receive placebo orally over a period of 7 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Niclosamide + Camostat — Niclosamide will be applied in combination with camostat.
  Other Names: Yomesan; Foipan
  Arms: Niclosamide + Camostat
Other: Placebo — Placebo to interventional drug
  Arms: Placebo

SUMMARY:
Niclosamide (2000 mg QD) and Camostate (600 mg QID) are expected to be safe and well-tolerated as a combination therapy and to show clinically beneficial for COVID-19 patients.

DETAILED DESCRIPTION:
Niclosamide is an approved drug for the treatment of intestinal worm infections that can potentially induce the process of autophagy and thus significantly limit viral replication in cells.

Camostat is approved in Japan for the treatment of chronic pancreatitis and reflux esophagitis. It has been shown to effectively block viral replication in a SARS-CoV-2 animal model.

Since the mechanisms of actions are different, it was hypothesized that a combination of both substances might have an additive or even synergistic effect in the treatment of patients with COVID-19.

This study is designed to investigate the safety, tolerability and preliminary efficacy of the treatment combination niclosamide and camostat in mild and moderately affected COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients in the age of 18 to 70 years
* Having a recent positive direct test for Sars-CoV-2
* Having mild or moderate COVID-19 symptoms with no indication for hospitalization due to SARS-CoV-2 infection (WHO Ordinal Scale 1-2)

Exclusion Criteria:

* Severe respiratory symptoms related to COVID-19 requiring oxygen or intensive care (high flow oxygen or mechanical ventilation or ECMO)
* Patients with preexisting pulmonary diseases requiring oxygen supply
* Patients with history of hypersensitivity to Camostat or Niclosamide or to any ingredients to any of the two drugs
* Patients with heart failure (NYHA III or NYHA IV)
* Patients with proven malignant tumor
* Patients diagnosed with influenza infection
* Pregnancy or breastfeeding
* Immunocompromised patients
* Creatinine clearance < 60 mL/min
* aspartate aminotransferase (AST) / alanine aminotransferase (ALT) > 2 times upper limit of normal (ULN)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Treatment emergent number of Adverse Events | 21 days
  All pathological and clinically significant findings in physical examinations, vital signs, 12-lead ECGs, oxygen saturation and safety lab including coagulation will be documented as adverse events. Adverse events will be reported on the basis of CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Witzenrath, Prof., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No